CLINICAL TRIAL: NCT00755950
Title: A Multicentre, Double-blind, Randomized, Placebo-controlled, Phase II/III Study to Evaluate the Safety and Efficacy of 280 mg and 420 mg Silymarin TID (Legalon® Capsules) Administered for Four Weeks in Subjects With Acute Viral Hepatitis With a Four Week Follow-up Period
Brief Title: Randomized Placebo-controlled Trial Evaluating the Safety and Efficacy of Silymarin Treatment in Patients With Acute Viral Hepatitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: MADAUS GmbH (Other); The Egyptian Company for Blood Transfusion Services (Other); Tanta Fever Hospital (Unknown); Banha Fever Hospital (Other); Alexandria University (Other)
Responsible Party: Principal Investigator, Samer S. El-Kamary, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HP-00042363; LE13K0.48
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Acute Hepatitis A; Acute Hepatitis B; Acute Hepatitis C; Acute Hepatitis E; Acute EBV Hepatitis; Acute CMV Hepatitis
Keywords: Acute; Hepatitis; Silymarin; Global Health
MeSH Terms: conditions — Hepatitis | interventions — Silymarin; milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 280 mg of Silymarin administered three times daily for 4 weeks; Vitamin B complex: B1:thiamine (1.3mg), B2:riboflavin (1.0mg) and B3: nicotinamide (16.5mg)
  Interventions: Dietary Supplement: Silymarin
- 3 (Placebo Comparator): Placebo: Lactose monohydrate; Vitamin B complex: B1:thiamine (1.3mg), B2:riboflavin (1.0mg) and B3: nicotinamide (16.5mg)
  Interventions: Other: Lactose monohydrate
- 2. (Experimental): 420 mg silymarin three times daily for four weeks; Vitamin B complex: B1:thiamine (1.3mg), B2:riboflavin (1.0mg) and B3: nicotinamide (16.5mg)
  Interventions: Dietary Supplement: Silymarin

INTERVENTIONS:
Dietary Supplement: Silymarin — 280 mg three times daily for four weeks
  Other Names: Legalon, Milk Thistle or St. Mary's Thistle
  Arms: 1
Dietary Supplement: Silymarin — 420 mg three times daily for four weeks
  Other Names: Legalon, Milk Thistle or St. Mary's Thistle
  Arms: 2.
Other: Lactose monohydrate — Lactose monohydrate 326.95 mg three times daily for four weeks
  Arms: 3

SUMMARY:
The purpose of this study is to assess whether two higher doses (280mg or 420mg three times daily)of silymarin therapy are safe and tolerable, and shorten the illness in patients with acute viral hepatitis compared to placebo.

DETAILED DESCRIPTION:
Currently, acute viral hepatitis (AVH) management is based on diet and rest and silymarin remains among the most popular herbs being used for treating viral hepatitis both in the U.S. and abroad. Although numerous randomized clinical trials have been conducted to assess the efficacy of silymarin on chronic hepatitis C, very few studies were done to assess the efficacy of silymarin in acute viral hepatitis. Among those, efficacy of silymarin has not been established. This could be attributed to the small number of studies conducted, small sample sizes, high drop out rates, and low doses of silymarin used. Therefore, it is justified to evaluate silymarin safety and efficacy using higher doses than previously studied in AVH.

Primary safety objective:

* To assess safety and tolerability of two silymarin doses in patients with AVH as determined by the number and percentage of subjects who develop Adverse Events in each group elicited by a questionnaire administered at specific visits and by hematology, blood chemistry and physical examinations.

Primary efficacy objective:

* To assess the percentage of subjects who normalize their total and direct bilirubin in each group.

Secondary Objective:

To assess the percentage of subjects in each group who:

* Normalize their liver enzymes, i.e. alanine aminotransferase (ALT), aspartate aminotransferase (AST) and inflammatory reactants, i.e. erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP).
* Resolve their clinical symptoms of AVH and return to baseline activity levels and quality of life (QOL) assessed by physical examinations and using a previously evaluated Arabic-translated SF-36 form adapted for use with patients with liver diseases.

To assess:

* Differences in silymarin response in different AVH etiologies (i.e. HAV, HBV, HCV, HEV) using subgroup analyses.

To compare:

* Progression of acute to chronic HCV infection in subjects with HCV-caused acute AVH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute viral hepatitis (<1 month) as manifested by a combination of the following symptoms: jaundice, dark-colored urine, light-colored stools, pruritus, pruritic red hives, fever, nausea, vomiting, anorexia, aversion to smoking and right upper abdominal discomfort, pain or feeling of pressure.
* Serum ALT level > 2.5 times the upper limit of normal.
* Albumin level >3.5 gm/dl
* Negative anti-HCV antibody
* Males and females >= 18 years of age.
* Subject has given written informed consent. If patient is between 18 and 21 years parents/legal guardian have/has also signed the informed consent form.
* The subject is able and willing to undertake all study-required procedures and has the ability to take oral medications.

Exclusion Criteria:

* Subjects < 18 years of age
* Pregnant or breastfeeding women
* Suspected hypersensitivity to silymarin or multivitamins
* Advanced liver disease (e.g. ascites, bleeding esophageal varices and hepatic encephalopathy)
* Chronic liver disease as cirrhosis
* Subjects with positive anti-HCV antibody
* Simultaneous elevation of bilirubin > 10 mg/dl along with an ALT level between 100 and 150 U/L
* Platelets count <150,000
* Subjects with morbid obesity i.e. a Body Mass Index (BMI) > 40
* Subjects with severe illness, e.g., multisystem failure, cancer or poorly controlled diabetes i.e. known diabetic with Hemoglobin A1C (HbA1C)>7%
* Obvious history of drug-induced acute hepatitis. A careful history of all medications, pesticide and other hepatotoxic exposures occurring within one month prior to symptom onset will be taken. If a patient is unaware of the name of the drugs, (s)he will be asked to bring it for inspection.
* Current use of Silymarin or recent use within past two weeks.
* Other conditions, which in the opinion of the investigators, makes the patient unsuitable for enrollment or could interfere with his/her participation in, and completion of, the protocol (e.g. severe mental illness)
* The subject is currently participating in any clinical trial (marketed product or otherwise), or has done so within 30 days or 5 half-lives (whichever is longer) prior to screening visit
* History or current drug or alcohol abuse
* Female patient with childbearing potential without negative pregnancy test
* Patient is known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and duration of Adverse Events | Four weeks after enrollment
Normalization of total (<1.0 mg/dl) and direct bilirubin (<0.3 mg/dl) | Four weeks after enrollment

SECONDARY OUTCOMES:
Normalization of ALT, AST, CRP and ESR | Four weeks after enrollment
Symptom resolution & return to normal physical activity | Eight weeks after enrollment
In AVH patients with specific etiologies resolution of clinical signs and symptoms | Eight weeks after enrollment
Persistence of acute HCV with progression to chronicity | Up to 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Samer El-Kamary, MD, MPH, Principal Investigator — University of Maryland, College Park; George T Strickland, MD, PhD,, Study Chair — University of Maryland, College Park; Mohamed Hashem, MD, Study Director — University of Maryland, College Park
Locations (3):
- Egypt (3):
  - Alexandria University Hospital, Alexandria, Alexandria Governorate
  - Tanta Fever Hospital, Tanta, Gharbeya Governorate
  - Banha Fever Hospital, Banhā, Kaluobeya Governorate